CLINICAL TRIAL: NCT04378335
Title: Assessment of Orality Disorders in Children With Food Allergies
Acronym: ALLERGORAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC19_0256
Record Dates: First submitted 2020-04-24; First posted 2020-05-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2020-04

CONDITIONS: Food Allergy in Children; 6 Years Old Maximum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm (Experimental): oral disorder
  Interventions: Other: completion of questionnaire

INTERVENTIONS:
Other: completion of questionnaire — parents have to complete 2 questionnaires: demographic questionnaire and Montréal questionnaire when they come on allergy consultation.

SUMMARY:
Orality disorders are frequent in child. There are complications like growth and psychomotor development disorders.

The aim is to estimate the prevalence of orality disorder for child with one or several food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Every child aged between 6 month and 6 years, with one or several food allergy and under the care of allergy unity of University Hospital of Angers
* obtention of informed consent

Exclusion Criteria:

* Child with allergy other than food
* poor understanding of french

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of orality disorder in children with food allergy | Enrollment

SECONDARY OUTCOMES:
Link between orality disorder and number of excluded food, time from excluded regimen, age of the beginning of diet diversification, breastfeeding and duration,status of the child in the family and demographic data. | Enrollment
  All data will be collected by a questionnaire established by Angers Hospital
Link between food allergies and orality disorder | Enrollment
  data will be collected by a questionnaire
Prevalence of dysphagia criteria | Enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No